CLINICAL TRIAL: NCT03162250
Title: A Phase IB, Randomized, Double-Blind, Placebo-Controlled, Multiple-Ascending Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of DSTA4637S in Patients With Staphylococcus Aureus Bacteremia Receiving Standard-of-Care Antibiotics
Brief Title: Study to Investigate the Safety, Tolerability, and Pharmacokinetics of DSTA4637S in Participants With Staphylococcus Aureus Bacteremia Receiving Standard-of-Care (SOC) Antibiotics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GV39131; 2016-001880-35 (EudraCT Number)
Record Dates: First submitted 2017-04-26; First posted 2017-05-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Bacteremia
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- DSTA4637S low dose level + SOC (Experimental): DSTA4637S low dose level intravenous (IV) infusion will be administered within 24 hours of randomization on Day 1 and then every 7 days up to 6 doses of study drug in addition to anti-staphylococcal SOC antibiotics.
  Interventions: Drug: DSTA4637S; Drug: SOC
- DSTA4637S intermediate dose level+ SOC (Experimental): DSTA4637S intermediate dose level IV infusion will be administered within 24 hours of randomization on Day 1 and then every 7 days up to 6 doses of study drug in addition to anti-staphylococcal SOC antibiotics.
  Interventions: Drug: DSTA4637S; Drug: SOC
- DSTA4637S high dose level+ SOC (Experimental): DSTA4637S high dose level IV infusion will be administered within 24 hours of randomization on Day 1 and then every 7 days up to 6 doses of study drug in addition to anti-staphylococcal SOC antibiotics.
  Interventions: Drug: DSTA4637S; Drug: SOC
- Placebo + SOC (Placebo Comparator): Placebo matched to DSTA4637S IV infusion will be administered within 24 hours of randomization on Day 1 and then every 7 days up to 6 doses of study drug in addition to anti-staphylococcal SOC antibiotics.
  Interventions: Drug: Placebo; Drug: SOC

INTERVENTIONS:
Drug: DSTA4637S — DSTA4637S will be administered as an IV infusion at 3 dose levels.
  Arms: DSTA4637S high dose level+ SOC; DSTA4637S intermediate dose level+ SOC; DSTA4637S low dose level + SOC
Drug: Placebo — Placebo matched to DSTA4637S IV infusion will be administered as specified.
  Arms: Placebo + SOC
Drug: SOC — Anti-staphylococcal SOC antibiotics dosage and duration of therapy will be based on relevant health-authority approved indications and local and national treatment guidelines.

SUMMARY:
This is a Phase Ib, randomized double-blind, placebo-controlled multiple-ascending dose study to investigate the safety, tolerability, and pharmacokinetics of multiple doses of DSTA4637S when given in addition to anti-staphylococcal SOC antibiotics to participants with methicillin-resistant staphylococcus aureus (MRSA) and methicillin-sensitive staphylococcus aureus (MSSA) bacteremia requiring at least 4 weeks of anti-staphylococcal SOC antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index greater than or equal (>/=) 18 to less than or equal to (</=) 40 kg/m^2
* At randomization, participants must have >/=1 blood culture or molecular diagnostic that is positive for Staphylococcal aureus (S. aureus) collected in the previous 120 hours
* In the investigator's judgment, an expected treatment duration for S. aureus intravenous infection with anti-staphylococcal SOC antibiotics >/= 4 weeks

Exclusion Criteria:

* The presence of an intravascular catheter that is not planned to be removed within 96 hours of study randomization
* S. aureus bacteremia associated with an intracardiac device and/or intravascular prosthetic material (including hemodialysis access graft)
* In the investigator's judgement, S. aureus bacteremia involving infection of a prosthetic joint or vertebral hardware
* In participants with cirrhosis, a Child-Pugh Score of Class B or C
* Known rifampicin-resistant S. aureus
* Anticipated receipt of a rifamycin class (excluding rifaxamin) antibiotic from Day 1 to study completion/discontinuation
* In the investigator's judgment, the need for emergent valve surgery at the time of randomization or a high likelihood of cardiac surgery within 3 days after randomization
* Polymicrobial bacteremia
* Participants with significant immune suppression
* Participants with evidence of liver disease
* History or presence of an abnormal electrocardiogram (ECG)
* Exposure to any biological therapy or investigational biological agent within 90 days prior to the screening evaluation or have received any other investigational treatment 30 days prior to the screening evaluation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) | Baseline up to approximately 156 Days

SECONDARY OUTCOMES:
Measure of Antibody-Conjugated 4-Dimethylamino Piperidino-Hydroxybenzoxazino Rifamycin (dmDNA31) measured by Plasma | Baseline up to approximately 156 Days
Measure of DSTA4637S Total Antibody measured by Serum | Baseline up to approximately 156 Days
Measure of Unconjugated dmDNA31 measured by Plasma | Baseline up to approximately 156 Days
Percentage of Participants With Anti-Therapeutic Antibodies (ATAs) to DSTA4637S | Baseline up to approximately 156 Days

CONTACTS AND LOCATIONS:
Locations (16):
- United States (4):
  - Los Angeles Biomedical Research Institute at Harbor-UCLA, Torrance, California
  - Henry Ford Health System, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Duke University Medical Center, Durham, North Carolina
- South Korea (4):
  - Chungnam National University Hospital, Daejeon
  - Gyeongsang National University Hospital, Gyeongsangnam-do
  - Asan Medical Center - Oncology, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (8):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital del Mar, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville